CLINICAL TRIAL: NCT06396455
Title: A Comparison Between Ultrasound Guided Suprascapular Nerve Block Versus Ultrasound Guided Interscalene Brachial Plexus Block on Respiratory Mechanics in Patients Undergoing Arthroscopic Shoulder Surgery: A Randomized Controlled Study
Brief Title: Ultrasound Guided Suprascapular Nerve Block Versus ISB Block in Arthroscopic Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ramy Mousa, Professor, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RC 16-1-2024
Record Dates: First submitted 2024-04-24; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Shoulder Surgery
Keywords: Anterior Suprascapular Nerve Block; Suprascapular Nerve Block

STUDY DESIGN:
Intervention Model Description: Group ISB (interscalene block group) received an ultrasound guided interscalene approach of brachial plexus plane block and group SSNB (suprascapular nerve block) received ultrasound guided suprascapular nerve block.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients, outcome assessors were blinded to the group allocation,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interscalene block group (Experimental): patients received an ultrasound guided interscalene approach of brachial plexus plane block
  Interventions: Procedure: interscalene block group
- suprascapular nerve block group (Experimental): patients received ultrasound guided suprascapular nerve block.
  Interventions: Procedure: Suprascapular nerve block group

INTERVENTIONS:
Procedure: interscalene block group — The ISB group scanning was done by linear ultrasound probe just below the level of the cricoid cartilage medial to the sternocleidomastoid muscle; the skin was disinfected, and the transducer was positioned in the transverse plane to identify the carotid artery. Once the artery was identified, the transducer was moved slightly laterally across the neck to identify the scalene muscles and the brachial plexus that is present between the anterior and middle scalene muscles. 3 ml lidocaine 1% was injected at puncture site The needle was then inserted in-plane toward the brachial plexus, in a lateral-to-medial direction. After a careful aspiration, 20 ml of bupivacaine 0.25% was injected.
  Other Names: Group ISB
  Arms: interscalene block group
Procedure: Suprascapular nerve block group — After cleaning the skin with an antiseptic solution, an ultrasound probe was put in sagittal orientation at the superior medial border of the scapula to identify the pleura and then moved laterally; when it was parallel to the spine of the scapula, the transducer was moved cephalad and the suprascapular fossa was identified, and then the transducer was moved lateral to locate the suprascapular notch. The suprascapular nerve was a round hyperechoic structure beneath the transverse scapular ligament in the scapular notch. 3 ml lidocaine 1% was injected at puncture site then the needle was inserted along the longitudinal axis of the ultrasound beam, and 10 ml of bupivacaine 0.25% was injected.
  Other Names: group SSNB
  Arms: suprascapular nerve block group

SUMMARY:
Diaphragmatic dysfunction can be detected as a decrease in forced vital capacity (FVC) and forced expiratory volume at 1 s (FEV1) on spirometry or as lower diaphragmatic excursion (DE) on US, the latter having become the gold standard in thoracic assessment.

DETAILED DESCRIPTION:
Severe intraoperative and postoperative pain associated with arthroscopic shoulder surgery has high incidence reaching up to 45%; it is often significant enough to interfere with initial recovery and rehabilitation.

Shoulder arthroscopy is becoming more common, representing the second most common Orthopedic surgery after knee arthroscopy . Interscalene brachial plexus block (ISB) is the gold standard analgesic technique for shoulder surgeries with success rates of 87% to 100%, but it also blocks the phrenic nerve (C3-C5).

Suprascapular nerve block via the anterior approach (SSB-A) is performed distally at the trunk/division level of the brachial plexus, thereby potentially sparing the phrenic nerve and minimising many adverse effects of ISB

ELIGIBILITY:
Inclusion Criteria:

* aged (18-65 years)
* American Society of Anesthesiologists (ASA) physical status I or II
* scheduled for elective arthroscopic shoulder surgery

Exclusion Criteria:

* pre-existing respiratory,
* cardiac, renal, neurological, or hepatic disease, neuropathy affecting brachial plexus
* contraindication to peripheral nerve block (e.g., coagulopathy),

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
visual analogue score | Postoperative pain was assessed using VAS at Postoperative care unit, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, and 24hours after block administration postoperatively
  The visual analogue score (VAS) was used (0 indicating no pain and 10 indicating worst unbearable pain) at rest and upon flexion for assessment of pain intensity upon arrival to the PACU

SECONDARY OUTCOMES:
Patient satisfaction | 24 hours postoperatively
  Patient satisfaction was evaluated using 5-point Likert scale) (1=extremely dissatisfied; 5=extremely satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Ramy Saleh, MD, Principal Investigator — Anesthesia and surgical ICU department, Faculty of Medicine, Benha University, Egypt
Locations (1):
- Benha University, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: No